CLINICAL TRIAL: NCT05058638
Title: Evaluation of Halitosis Using a Multi-Mineral Approach (Aquamin®)
Brief Title: Effectiveness of Aquamin® in Mitigating Halitosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Muhammad N Aslam, MD, Associate Research Scientist, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00156676 Halitosis substudy
Record Dates: First submitted 2021-09-16; First posted 2021-09-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Halitosis
Keywords: Aquamin®
MeSH Terms: conditions — Halitosis | interventions — Aquamin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aquamin® (Experimental)
  Interventions: Drug: Aquamin

INTERVENTIONS:
Drug: Aquamin — Participants will take a 90-day supply of Aquamin®, 4 capsules per day; 2 to be taken in the morning and 2 in the evening (containing approximately 800 mg calcium/day).
  Other Names: Nutritional

SUMMARY:
The purpose of this study is to assess whether Aquamin®, a multi-mineral natural product from red marine algae, can help reduce halitosis when taken for 90 days.

DETAILED DESCRIPTION:
This is a sub-study to the ongoing clinical trial entitled: Aquamin®, a multi-mineral natural product from red marine algae, as an adjuvant intervention for mild ulcerative colitis and ulcerative colitis in remission (HUM00156676) NCT# NCT03869905.

However, the Food and Drug Administration (FDA) indicated that no Investigational New Drug Application (IND) was required.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to give written informed consent
* Willing to follow study procedures of no eating, drinking, toothbrushing, smoking or using mouth rinse 60 minutes before study visits
* Willing to not scrape their tongue with a toothbrush, oral hygiene aid, or other utensil during the study participation
* Periodontally stable
* Self-reported halitosis
* A negative pregnancy test for pre-menopausal women with intact female reproductive organs, and subject must agree to use appropriate birth control over the study period.

Exclusion Criteria:

* Pregnant or lactating women
* Participating in any other interventional trials using an investigational drug
* Diagnosed with any stomach or intestinal bleeding disorders (gastrointestinal bleeding from gastric or duodenal ulcers, or gastrin secreting tumors) or active gastric / duodenal ulcers - peptic ulcer disease (in last 3 months) or with severe symptoms of ulcerative colitis or Crohn's disease
* Any gastrointestinal or colonic malignancy- Kidney disease, including kidney "stones" or hypercalcemia
* Coagulopathy/hereditary hemorrhagic disorders/or receiving therapeutic doses of Coumadin or heparin
* Presence of one or more cavitated carious lesions, untreated dental abscesses (endodontic or periodontal), untreated periodontitis (gum disease), or oral pathologies that may contribute to oral malodor (e.g., candidiasis, erosive gingival conditions)
* Taking any of the following within 30 days (will be eligible after completing 30 days of wash out period):

Calcium; Vitamin D, including multivitamins that have low amounts of calcium/Vitamin D supplements; Oral steroids; Non-steroidal anti-inflammatory medications (NSAIDS); Antibiotics.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Halitosis Associated Life-quality Test (HALT) questionnaire (modified) | 90 days (post-intervention)
  Following the intervention, participants will answer questions regarding if their bad breath has improved over the course of the study compared to the starting point. The scores will be from 0 (no issue) - 5 (worst possible issue) for each question.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad N Aslam, Principal Investigator — University of Michigan; Janet Kinney, Study Director — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No